CLINICAL TRIAL: NCT05890378
Title: Integrated Livestock Management for Nutrition in Children Under Five Years of Age
Brief Title: Integrated Livestock Management for Nutrition in Children Under Five Years of Age in Chad
Status: Not yet recruiting | Type: Observational
Sponsor: Tufts University (Other)
Collaborators: Food and Agriculture Organization of the United Nations (Unknown)
Responsible Party: Sponsor
Other Study IDs: Marshak-FAO-Chad
Record Dates: First submitted 2023-05-25; First posted 2023-06-06 (Actual); Last update posted 2023-06-07 (Actual); Status verified 2023-06

CONDITIONS: Malnutrition, Child
Keywords: malnutrition
MeSH Terms: conditions — Child Nutrition Disorders; Malnutrition

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — fecal matter
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cohort by Water Source: Using existing secondary data available on the research communities as well as qualitative inquiry, we will purposefully select 40 water sources for the water analysis across from the communities selected for the implementation research (up to 30 communities with a maximum of 5 water sources per community). The selection of water sources will be stratified by type of water sourceand near the route for long-term animal migration. For each water source, we will aim to have a water sample collected at all water sources twice a day (morning and later afternoon) once a week for four weeks, varying the day of the week. Thus, we will collect a total of 320 water samples in the course of four weeks at the end of the dry season before the rains start.
  Interventions: Other: Testing water

INTERVENTIONS:
Other: Testing water — Using existing secondary data available on the research communities as well as qualitative inquiry, we will purposefully select 40 water sources for the water analysis across from the communities selected for the implementation research (up to 30 communities with a maximum of 5 water sources per community). The selection of water sources will be stratified by type of water sourceand near the route for long-term animal migration. For each water source, we will aim to have a water sample collected at all water sources twice a day (morning and later afternoon) once a week for four weeks, varying the day of the week. Thus, we will collect a total of 320 water samples in the course of four weeks at the end of the dry season before the rains start.

SUMMARY:
The main objective of this study is to determine the effectiveness of a livestock management intervention, with considerations for animal food security, water contamination from animals, and nutrition counseling, in reducing the risk of acute malnutrition among children under the age of 5 years in Kanem and Bahr El Ghazel (BeG) in Chad.

DETAILED DESCRIPTION:
The main objective of this study is to determine the effectiveness of a livestock management intervention, with considerations for animal food security, water contamination from animals, and nutrition counseling, in reducing the risk of acute malnutrition among children under the age of 5 years in Kanem and Bahr El Ghazel (BeG) in Chad. To get at this objective we will be comparing across four study arms: 1) fodder provision, 2) water management/treatment, 3) combination of fodder and water management/treatment and 4) a control. All four arms will receive nutrition counseling, animal vaccination, and animal deworming.

Specifically, the study aims to answer the following research questions in the implementation research:

1. Does provision of animal feed and nutrition counseling lead to a reduction in child acute malnutrition of children under five?
2. Does messaging pulling on existing local strategies to improve protected water access for animals and humans, provision of a chlorine dispenser, and nutrition counseling lead to a reduction in child acute malnutrition of children under five?
3. Does provision of animal feed, nutrition counseling, in combination with messaging pulling on existing local strategies to improve protected water access for animals and humans lead to a reduction in child acute malnutrition of children under five?

In preparation for the implementation of the intervention, we will conduct formative research to better contextualize the interventions and data collection. The formative research will seek to answer the following research questions.

1. What is the water quality of and practices around different types of unimproved water sources?
2. Which water sources are used by households, and what is their distance from the community?
3. What zoonotic pathogens are present in animal and human fecal matter, and in milk?
4. What is the highest acceptable (using the flavor rating assessment method - Table 5) concentration of chlorine to provide safe water for users?

The study will be done in a phased approach:

* Year 1: formative research
* Year 2: impact evaluation
* Year 3: sustainability study

ELIGIBILITY:
Inclusion Criteria:

* Communities selected for the research have to be near a seasonal river
* Households (within those communities) have to have at least one child between the ages of 6 and 59 months.
* Households (within those communities) have to have at least one Tropical Livestock Unit (TLU) of livestock. One TLU is equivalent to either one cow, one camel, 10 goats or 10 sheep.
* Within those households, we will interview the female caretaker
* Anthropometry data will be collected from children 6-59 months and the female caretaker

Exclusion Criteria:

* lack of children under 5 years of age and/or a required livestock unit

Ages: 6 Months to 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Although the final target for many nutrition messages will be women with young children, their ability to carry out promoted practices depends on the influence and control of a range of actors. Likewise, both men and women in households with livestock make decisions that affect resources provided to milking animals and access to milk - and these individuals are affected by a range of other actors in the community.
Sampling Method: Non-Probability Sample
Enrollment: 15000 (Estimated)
Dates: Start 2023-07 (Estimated); Primary Completion 2026-02 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Water Quality | 2023-2026
  Water quality: total coliform and E. coli

IPD SHARING:
Plan to Share IPD: No